CLINICAL TRIAL: NCT02994238
Title: iTRACC (Improving Technology-Assisted Recording of Asthma Control in Children)
Acronym: iTRACC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Deneen Vojta (Industry)
Collaborators: Northwestern University (Other)
Responsible Party: Sponsor-Investigator, Dr. Deneen Vojta, Executive Vice President, Research and Development, UnitedHealth Group, UnitedHealth Group
Organization: UnitedHealth Group (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB 2016-698
Record Dates: First submitted 2016-11-04; First posted 2016-12-15 (Estimated); Results first posted 2021-08-24 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The intervention group will have the full Remote Health Management Sensor Platform. Research staff will review uploaded sensor data on a daily basis. If participants are enrolled into the control group, they will only receive Standard Asthma Education. The Standard Asthma Education follows the National Asthma Education and Prevention Program (NAEPP) guidelines for asthma management. This will include the following topics: 1. Explanation of symptoms; 2. Asthma triggers (description and how to avoid them); 3. Using medications (how to use prescribed asthma medications, the difference between controller medications and rescue inhalers, how to use a spacer, how to use a mask); and 4. Managing asthma control (purpose of asthma control test, asthma action plan, how to use a peak flow meter).
  Interventions: Device: Remote Health Management Sensor Platform
- Control (No Intervention): The control group will receive only standardized education.

INTERVENTIONS:
Device: Remote Health Management Sensor Platform — The Propeller sensor monitors the use of inhaled medications, capturing the date, time, and number of uses. The sensor then transmits this information using Bluetooth to a paired smart phone or hub. Data can be uploaded to the caregiver's smart phone and to the patient's web portal, which their healthcare team will have access to help overall management.
  Other Names: Reciprocal Labs; Propeller Health Systems
  Arms: Intervention

SUMMARY:
The goal of this study is to determine whether a sensor-enabled, clinically integrated, mobile health asthma program can improve asthma outcomes among 4-17 year old children with moderate-to-severe asthma.

DETAILED DESCRIPTION:
Primary Aims:

* Assess whether asthma control in patients enrolled in the intervention arm improved in comparison to the control arm through the (ACT) measurement tool.
* Assess healthcare utilization (asthma-related ED visits and hospitalizations, asthma-related oral corticosteroid use) obtained through electronic medical record and parent report.

Secondary Aims:

Investigators will use parent-report surveys of the following psycho-social outcome measures:

* Days missed from school due to asthma; 2) pediatric asthma-related quality of life (PACQLQ); and 3) Parental Asthma Management Self-Efficacy (PAMSE).
* Enhance parental management through improved inhaler use. The investigators will use the Propeller Sensor Platform (referenced as Remote Health Management Platform) to allow parents to track their child's ICS and SABA inhaler use daily. The Platform also will have specific educational messaging to help parents and their children achieve adherence to their prescribed plan. This constant feedback and reinforcement may lead to improved asthma control therefore reducing frequency and severity of asthma exacerbations. The investigators will also be assessing the factors associated with the feasibility and sustainability of the Propeller Sensor Platform by observing trends in utilization. Utilization and drop-off will be measured by monitoring use of the inhalers and periodic surveys of families.
* Improve management by the healthcare team. The investigators will use the Remote Health Management Platform to integrate inhaler use data into a web portal that the physician's office can access. Through the development of this interface, the Propeller Sensor Platform will be able to provide inhaler use feedback to healthcare teams.

Types of feedback:

* Emergency Management: data on inhaled corticosteroids (ICS) and short-acting beta-agonist (SABA) use
* Long-term Management: data on ICS and SABA use. This interface will include data on both ICS and SABA inhaler use. The interface will also have flags to notify the office of under or overuse of inhalers, with a protocol in place to reach out to patients. The investigators will also be assessing the factors associated with the feasibility and sustainability of the Remote Health Management Platform by the healthcare team. This will be done by weekly contact with the healthcare team, rapid cycle improvement of the web portal, and written assessments.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking parents
* Children 4-<17 years of age. Using both NHLBI (National Heart, Lung, and Blood Institute) guidelines and based off of a physician expert panel, the research team has limited the ages to 4-<17 years old. It has been shown to be difficult to properly diagnose individuals less than 4 years of age with asthma. Usually, they are diagnosed with reactive airway disease or bronchial virus. Individuals <17 years old was the oldest group because investigators wanted to avoid adolescence and make sure that parents have an active role in the health management of the child.
* Moderate or severe persistent asthma, defined by the National Heart, Lung, and Blood Institute. This will be done by a physician-trained research assistant who will be able to identify potential participants prior to recruitment.
* At least one asthma exacerbations that required a course of oral corticosteroids in the past year
* Prescription and utilization of an ICS inhaler for at least the past year.
* Who are seen at: Clark and Deming Resident Clinic, Lurie Children's Pulmonary Clinic, Lurie Children's Uptown Clinic, Chicago Family Asthma and Allergy Clinic or Children's Healthcare Associates

Exclusion Criteria:

* Non-English speaking parents/families
* Patients seen in the hospital who receive primary care outside of the study's clinics
* Children with any comorbid conditions, which interfere with appropriate assessment of asthma symptoms: Chronic Lung Disease, Broncho-Pulmonary Dysplasia, Cystic Fibrosis, Pulmonary Hypertension, Interstitial Lung Disease, Immunodeficiency, Bronchiectasis, Primary Ciliary Dyskinesia, Chronic Respiratory Insufficiency, Neuromuscular Weakness, Sickle Cell Lung Disease, Restrictive Lung Disease, and Tracheostomy or Ventilator-dependence
* Child-patients who are participating in any other research studies that would interfere with our ability to use and track the inhaler sensor

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 252 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12-31 (Actual)

REFERENCES:
- [Derived] Gupta RS, Fierstein JL, Boon KL, Kanaley MK, Bozen A, Kan K, Vojta D, Warren CM. Sensor-Based Electronic Monitoring for Asthma: A Randomized Controlled Trial. Pediatrics. 2021 Jan;147(1):e20201330. doi: 10.1542/peds.2020-1330. PMID 33386336

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 125 | 127
Completed | 125 | 127
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 125 | 127 | 252
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 125 | 127 | 252
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.3 (3.2) | 9.2 (3.5) | 9.2 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: some patients did not choose to identify sex as either male or female
  Participants
    number analyzed (Participants) | 114 | 125 | 239
    Female | 44 | 39 | 83
    Male | 70 | 86 | 156
Race/Ethnicity, Customized [Number; unit: Percentage of participants]
  Non-Hispanic/White % | 24.0 | 23.6 | 47.6
  Non-Hispanic/Black % | 23.2 | 33.1 | 56.3
  Hispanic % | 40.0 | 28.4 | 68.4
  Other Race/Ethnicity % | 7.2 | 7.8 | 15.0
  No Data % | 5.6 | 7.1 | 12.7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 125 | 127 | 252
Insurance Type [Number; unit: Percentage of participants]
  Private Insurance % | 40 | 43.3 | 42.8
  Public Insurance % | 59.2 | 56.7 | 57.2
ACT Score [Mean (Standard Deviation); unit: units on a scale] — Investigators will use the children's Asthma Control Test completed by the caregiver or parent to report child's asthma control. The ACT is a 5 item scale, with a 4-week recall (on symptoms and daily functioning) ACT assesses the frequency of shortness of breath and general asthma symptoms, use of rescue medications, the effect of asthma on daily functioning, and overall self-assessment of asthma control via item-specific response options ranging from 1-5. Total ACT scores range from 5 (poorly controlled asthma, to 25 (well controlled asthma).
  units on a scale | 18.8 (4.5) | 19.6 (3.8) | 19.2 (4.2)
PACQLQ [Mean (Standard Deviation); unit: units on a scale] — The Pediatric Asthma Caregiver Quality of Life (QOL) Questionnaire was administered. This scale is a self-administered instrument, which includes 13 items (4 concern activity limitations and 9 concern emotional function). Responses to each item of the PACQLQ are given on a seven-point scale, ranging from 1 to 7, with the higher scores indicating less impairment. A total average score was calculated to reflect Pediatric Asthma Caregiver Quality of Life, which also ranged from 1-7.
  units on a scale | 5.7 (1.3) | 5.8 (1.1) | 5.8 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Asthma Control Test (ACT)
Description: Investigators will use the children's Asthma Control Test completed by the caregiver or parent to report child's asthma control. The ACT is a 5 item scale, with a 4-week recall (on symptoms and daily functioning) ACT assesses the frequency of shortness of breath and general asthma symptoms, use of rescue medications, the effect of asthma on daily functioning, and overall self-assessment of asthma control via item-specific response options ranging from 1-5. Total ACT scores range from 5 (poorly controlled asthma, to 25 (well controlled asthma).
Time Frame: 12 month follow-up assessment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 125 | 127
units on a scale | 21.8 (.4) | 19.9 (.4)

2. Primary Outcome: Frequency of Urgent Health Utilization
Description: Number of Asthma-related ED visits during the 12 month study period
Time Frame: the 12 month study period
Measure: Mean (Standard Error); unit: events (asthma-related ED visits)
Arm/Group | Intervention | Control
Number analyzed (Participants) | 125 | 127
events (asthma-related ED visits) | 1.0 (.1) | .6 (.1)

3. Primary Outcome: 12 Month Rate of Medication Use
Description: Number of oral corticosteroid prescriptions obtained from the electronic medical record and parent/caregiver report
Time Frame: Over a 12 month study period
Measure: Mean (Standard Error); unit: OCS Prescriptions
Arm/Group | Intervention | Control
Number analyzed (Participants) | 125 | 127
OCS Prescriptions | 1.3 (.2) | .9 (.2)

4. Secondary Outcome: Pediatric Asthma Caregiver Quality of Life (QOL) Questionnaire
Description: The Pediatric Asthma Caregiver Quality of Life (QOL) Questionnaire was administered. This scale is a self-administered instrument, which includes 13 items (4 concern activity limitations and 9 concern emotional function). Responses to each item of the PACQLQ are given on a seven-point scale, ranging from 1 to 7, with the higher scores indicating less impairment. A total average score was calculated to reflect Pediatric Asthma Caregiver Quality of Life, which also ranged from 1-7.
Time Frame: 12 month study follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 125 | 127
units on a scale | 6.3 (1.0) | 6.0 (1.4)

5. Primary Outcome: Frequency of Asthma-related Hospitalizations
Description: Number of Asthma-related Hospitalizations during the 12 month study period
Time Frame: the 12 month study period
Measure: Mean (Standard Error); unit: Events (Asthma-related Hospitalizations)
Arm/Group | Intervention | Control
Number analyzed (Participants) | 125 | 127
Events (Asthma-related Hospitalizations) | .4 (.1) | .1 (.06)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/125 | 0/127
Serious Adverse Events (participants affected / at risk) | 0/125 | 0/127
Other Adverse Events (participants affected / at risk) | 0/125 | 0/127

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/38/NCT02994238/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/38/NCT02994238/SAP_001.pdf